CLINICAL TRIAL: NCT05938608
Title: An Open-Label Pharmacokinetic Study to Evaluate the Bioavailability of Oral Primaquine and the Pharmacokinetics of Carboxyprimaquine in Healthy Adult Subjects
Brief Title: A Study to Assess the Availability of Oral Primaquine and Its Inert Metabolite, Carboxyprimaquine, in the Body
Acronym: PQcPQ
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study team's decision to withdraw the study.
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAL22006
Record Dates: First submitted 2023-06-22; First posted 2023-07-10 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Pharmacokinetic
Keywords: Primaquine; Carboxyprimaquine
MeSH Terms: interventions — Primaquine; 8-(3-carboxy-1-methylpropylamino)-6-methoxyquinoline

STUDY DESIGN:
Intervention Model Description: This is an open-label pharmacokinetic study in 20 healthy adult subjects. Subjects will be admitted in the hospital and will receive 3 regimens of primaquine and its metabolite. Every subject will have 1 screening and 3 admissions in the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regimen 1 (Oral primaquine), 2(IV primaquine phosphate), 3(IV carboxyprimaquine) (Experimental): Regimen 1 (Oral primaquine): Primaquine 15 mg base orally once
  Regimen 2 (IV primaquine phosphate): Primaquine 7.5 mg base in normal saline 500 mL infused over 30 minutes intravenously
  Regimen 3 (IV carboxyprimaquine): Carboxyprimaquine 7.93 mg base in normal saline 500 mL infused over 30 minutes intravenously
  Interventions: Drug: Regimen 1 (Oral primaquine); Drug: Regimen 2 (IV primaquine phosphate); Drug: Regimen 3 (IV carboxyprimaquine)

INTERVENTIONS:
Drug: Regimen 1 (Oral primaquine) — Primaquine 15 mg base orally once
Drug: Regimen 2 (IV primaquine phosphate) — Primaquine 7.5 mg base in normal saline 500 mL infused over 30 minutes intravenously
Drug: Regimen 3 (IV carboxyprimaquine) — Carboxyprimaquine 7.93 mg base in normal saline 500 mL infused over 30 minutes intravenously

SUMMARY:
An open-label pharmacokinetic study. This study will enroll 20 healthy adult subjects (10 males and 10 females aged 18-60 years) at the Clinical Therapeutics Unit or inpatient ward, Faculty of Tropical Medicine, Mahidol University, Thailand.

The investigator propose to conduct a definitive bioavailability and pharmacokinetic study in healthy adult volunteers, both male and female, with normal CYP2D6 genotypes to assess oral primaquine bioavailability by the administration of intravenous and oral primaquine on different days and calculate the proportion of drug converted to its inactive metabolite, carboxyprimaquine, in order to estimate the proportion of its active metabolites. The intravenous injection of the known amount of carboxyprimaquine will allow the calculation of carboxyprimaquine's volume of distribution.

DETAILED DESCRIPTION:
This study will enroll 20 healthy adult subjects (10 males and 10 females aged 18-60 years).

Subjects will be admitted in the hospital and will receive 3 regimens of primaquine and its metabolite as described below. Every subject will have 1 screening and 3 admissions in the hospital.

Regimen 1: Primaquine 15 mg base orally once

Regimen 2: Primaquine 7.5 mg base in normal saline 500 mL infused over 30 minutes intravenously

Regimen 3: Carboxyprimaquine 7.93 mg base in normal saline 500 mL infused over 30 minutes intravenously

Washout period will be at least 2 weeks between each regimen.

The pharmacokinetic blood samples, 2 mL, will be collected at the scheduled times relative to when the subject was dosed for each regimens as follow.

Regimen 1: 16 blood samples collected from day 1 at 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours post-dose, day 1 at 24 hours post-dose, day 2 at 48 hours post-dose and only 1 sampling at any time on day 3, 5 and 7.

Regimen 2 and 3: 17 blood samples collected from day 1 at 0 (pre-dose), 0.25 (during), 0.5 (immediately after), 0.75, 1, 2, 3, 4, 6, 8, 10, 12 hours post-dose, day 1 at 24 hours post-dose, day 2 at 48 hours post-dose and only 1 sampling at any time on day 3, 5 and 7.

Plasma samples will be assayed by a validated Liquid Chromatography-Mass Spectrometer (LCMS/MS) method developed at Mahidol Oxford Tropical Medicine Research Unit (MORU), which is specific for the determination of primaquine and its metabolite, carboxyprimaquine.

Individual concentration-time data will be evaluated using a non-compartmental analysis approach. Pharmacokinetic parameters (i.e. Area under the concentration-time curve (AUC0-LAST, AUC0-∞), Maximum concentration (CMAX), Time to maximum concentration (TMAX), elimination clearance (CL/F), apparent volume of distribution (VD/F), and terminal elimination half-life (t1/2)) will be described using means (SD or 95% CI) and medians (range) as appropriate. Bioavailability of oral primaquine will be calculate based on the dose-normalised exposure (AUC0-LAST and AUC0-∞) to primaquine after oral and intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as judged by a responsible physician with no significant abnormality identified on a medical evaluation including medical history and physical examination.
2. Male or female aged between 18 years to 60 years.
3. A female is eligible to enter and participate in this study if she is:

   • of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy

   OR

   • postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 milli-international units per milliliter (mIU/mL) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy

   OR

   • of childbearing potential, has a negative serum pregnancy test at screening and urine pregnancy test prior to start the study drug in each period, and agrees to abstain from sexual intercourse or use effective contraceptive methods (e.g., intrauterine device, tubal ligation or female barrier method with spermicide except hormonal contraceptive) during the study until completion of the follow-up procedures
4. Willingness and ability to comply with the study protocol for the duration of the trial.
5. Subject is willing and able to give written informed consent for full participation in the study

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. Known to have any clinically significant disease or to have a clinically significant disease or disorder at this screening time
3. Donated more than 300 mL of whole blood within the previous 3 months
4. Non-smokers and non-tobacco user (i.e. having no past history of smoking and tobacco consuming for at least 3 months prior to study)
5. Consume alcohol or other alcohol containing products within 48 hours prior to the first dose of study drug and throughout the study
6. History or evidence of alcohol or substance abuse or dependence within 6 months before and throughout the study
7. Consume grapefruit and grapefruit containing products within 7 days prior to the first dose of study drug and throughout the study
8. Use of prescription drugs including but not limited to drugs with antimalarial activities and any drug contraindicated with the investigational drugs e.g. quinacrine, mefloquine or non-prescription drug, including, vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and for the duration of the trial including follow-up will be prohibited
9. Have taken part in research involving an investigational drug within the past 8 weeks
10. Use of medications known to have a potentially clinically significant interaction with primaquine
11. History of allergy to primaquine
12. Hb < 11 g/dL
13. Having malaria infection
14. Abnormal CYP2D6 genotype
15. Glucose-6-phosphate dehydrogenase (G6PD) deficiency by screening test
16. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 1.5 times the upper limit of normal (ULN)
17. A serum creatinine (Scr) above the upper limit of normal (> 1.2 mg/dL) and estimated glomerular filtration rate (eGFR) < 70 mL/min/1.73 m2
18. Methaemoglobin (MetHb) level > 3% determined by oximetry
19. Positive for HIV-1, Hepatitis B or C virus infection
20. Subject who is likely to be unable to follow with the study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC0-∞) of oral and intravenous primaquine. | Approximately 3 months
Area under the concentration-time curve (AUC0-last) of oral and intravenous primaquine. | Approximately 3 months
Area under the concentration-time curve (AUC0-∞) of primaquine and carboxyprimaquine | Approximately 3 months
Area under the concentration-time curve (AUC0-last) of primaquine and carboxyprimaquine | Approximately 3 months
Maximum concentration (Cmax) of primaquine and carboxyprimaquine | Approximately 3 months
Elimination clearance (CL/F) of primaquine and carboxyprimaquine | Approximately 3 months
Terminal elimination half-life (t1/2) of primaquine and carboxyprimaquine | Approximately 3 months
Apparent volume of distribution (Vd) of primaquine and carboxyprimaquine | Approximately 3 months

SECONDARY OUTCOMES:
The characteristics of genetic polymorphisms of potential enzymes involved in drug metabolism in the case of unusual metabolizer | Approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Borimas Hanboonkunupakarn, Asst. Prof, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
With subject's consent, subject's clinical data and results from blood analyses stored in our database may be shared with other researchers to use in the future. However, the other researchers will not be given any information that could identify the subject.
Access Criteria: Access to study data will be provided following the MORU data sharing policy.
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing